CLINICAL TRIAL: NCT00839527
Title: A Randomized, Double-blind, Placebo and Active-Controlled, Parallel-group, Multicenter Study to Determine the Efficacy and Safety of Albiglutide Administered in Combination With Metformin and Glimepiride Compared With Metformin Plus Glimepiride and Placebo and With Metformin Plus Glimepiride and Pioglitazone in Subjects With Type 2 Diabetes Mellitus
Brief Title: A Study to Determine the Safety and Efficacy of Albiglutide in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 112757
Record Dates: First submitted 2009-02-05; First posted 2009-02-09 (Estimated); Results first posted 2014-07-01 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — rGLP-1 protein; Metformin; glimepiride; Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- metformin + glimepiride + pioglitazone + albiglutide placebo (Active Comparator): Metformin + glimepiride + pioglitazone + matching albiglutide placebo
  Interventions: Drug: placebo to match albiglutide; Drug: metformin; Drug: glimepiride; Drug: pioglitazone
- metformin + glimepiride + pioglitazone placebo + albiglutide (Experimental): Metformin + open-label glimepiride + pioglitazone matching placebo + albiglutide
  Interventions: Biological: albiglutide; Drug: metformin; Drug: glimepiride; Drug: placebo to match pioglitazone
- met + glimepiride + pioglitazone placebo + albiglutide placebo (Active Comparator): metformin + open-label glimepiride + pioglitazone placebo + albiglutide placebo
  Interventions: Drug: placebo to match albiglutide; Drug: metformin; Drug: glimepiride; Drug: placebo to match pioglitazone

INTERVENTIONS:
Drug: placebo to match albiglutide — albiglutide matching placebo weekly subcutaneous injection
  Arms: met + glimepiride + pioglitazone placebo + albiglutide placebo; metformin + glimepiride + pioglitazone + albiglutide placebo
Biological: albiglutide — albiglutide weekly subcutaneous injection
  Arms: metformin + glimepiride + pioglitazone placebo + albiglutide
Drug: metformin — metformin
Drug: glimepiride — glimepiride
Drug: pioglitazone — pioglitazone
  Arms: metformin + glimepiride + pioglitazone + albiglutide placebo
Drug: placebo to match pioglitazone — pioglitazone matching placebo
  Arms: met + glimepiride + pioglitazone placebo + albiglutide placebo; metformin + glimepiride + pioglitazone placebo + albiglutide

SUMMARY:
The purpose of this study is to determine the safety and efficacy of albiglutide in subjects with type 2 diabetes

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes
* BMI 20-45kg/m2 inclusive

Exclusion Criteria:

* females who are pregnant, lactating, or less than 6 weeks post-partum
* current symptomatic heart failure (NYHA Class II-IV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 685 (Actual)
Dates: Start 2009-02; Primary Completion 2012-01 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (294):
- United States (260):
  - GSK Investigational Site, Alabaster, Alabama
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Dothan, Alabama
  - GSK Investigational Site, Mobile, Alabama
  - GSK Investigational Site, Tuscaloosa, Alabama
  - GSK Investigational Site, Chandler, Arizona
  - GSK Investigational Site, Gilbert, Arizona
  - GSK Investigational Site, Green Valley, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Bull Shoals, Arkansas
  - GSK Investigational Site, Harrisburg, Arkansas
  - GSK Investigational Site, Hot Springs, Arkansas
  - GSK Investigational Site, Jonesboro, Arkansas
  - GSK Investigational Site, Searcy, Arkansas
  - GSK Investigational Site, Buena Park, California
  - GSK Investigational Site, Chino, California
  - GSK Investigational Site, Chula Vista, California
  - GSK Investigational Site, Commerce, California
  - GSK Investigational Site, Escondido, California
  - GSK Investigational Site, Foothill Ranch, California
  - GSK Investigational Site, Fountain Valley, California
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Fullerton, California
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Indio, California
  - GSK Investigational Site, La Jolla, California
  - GSK Investigational Site, Lakewood, California
  - GSK Investigational Site, Loma Linda, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Alamitos, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Mission Viejo, California
  - GSK Investigational Site, Northridge, California
  - GSK Investigational Site, Palm Desert, California
  - GSK Investigational Site, Palm Springs, California
  - GSK Investigational Site, Pasadena, California
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Santa Ana, California
  - GSK Investigational Site, Satna Monica, California
  - GSK Investigational Site, Spring Valley, California
  - GSK Investigational Site, Tarzana, California
  - GSK Investigational Site, Tustin, California
  - GSK Investigational Site, Victorville, California
  - GSK Investigational Site, Walnut Creek, California
  - GSK Investigational Site, West Hills, California
  - GSK Investigational Site, Arvada, Colorado
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, New Britain, Connecticut
  - GSK Investigational Site, Trumbull, Connecticut
  - GSK Investigational Site, Waterbury, Connecticut
  - GSK Investigational Site, Middletown, Delaware
  - GSK Investigational Site, Boynton Beach, Florida
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, Cocoa, Florida
  - GSK Investigational Site, Cutler Bay, Florida
  - GSK Investigational Site, Deerfield Beach, Florida
  - GSK Investigational Site, Delray Beach, Florida
  - GSK Investigational Site, Edgewater, Florida
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Gainesville, Florida
  - GSK Investigational Site, Hallandale, Florida
  - GSK Investigational Site, Hialeah, Florida
  - GSK Investigational Site, Hollywood, Florida
  - GSK Investigational Site, Lauderdale Lakes, Florida
  - GSK Investigational Site, Marianna, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, North Miami, Florida
  - GSK Investigational Site, Ocala, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Ormond Beach, Florida
  - GSK Investigational Site, Oviedo, Florida
  - GSK Investigational Site, Panama City, Florida
  - GSK Investigational Site, Pembroke Pines, Florida
  - GSK Investigational Site, Plantation, Florida
  - GSK Investigational Site, Ponte Verda, Florida
  - GSK Investigational Site, Saint Cloud, Florida
  - GSK Investigational Site, St. Petersburg, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Blue Ridge, Georgia
  - GSK Investigational Site, Columbus, Georgia
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Savannah, Georgia
  - GSK Investigational Site, Snellville, Georgia
  - GSK Investigational Site, Stone Mountain, Georgia
  - GSK Investigational Site, Tucker, Georgia
  - GSK Investigational Site, Honolulu, Hawaii
  - GSK Investigational Site, Boise, Idaho
  - GSK Investigational Site, Idaho Falls, Idaho
  - GSK Investigational Site, Aurora, Illinois
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Evergreen Park, Illinois
  - GSK Investigational Site, Gurnee, Illinois
  - GSK Investigational Site, La Grange, Illinois
  - GSK Investigational Site, Naperville, Illinois
  - GSK Investigational Site, Peoria, Illinois
  - GSK Investigational Site, Avon, Indiana
  - GSK Investigational Site, Evansville, Indiana
  - GSK Investigational Site, Fishers, Indiana
  - GSK Investigational Site, La Porte, Indiana
  - GSK Investigational Site, Lafayette, Indiana
  - GSK Investigational Site, South Bend, Indiana
  - GSK Investigational Site, Council Bluffs, Iowa
  - GSK Investigational Site, Des Moines, Iowa
  - GSK Investigational Site, Dubuque, Iowa
  - GSK Investigational Site, Iowa City, Iowa
  - GSK Investigational Site, Waterloo, Iowa
  - GSK Investigational Site, Arkansas City, Kansas
  - GSK Investigational Site, Mission, Kansas
  - GSK Investigational Site, Newton, Kansas
  - GSK Investigational Site, Overland Park, Kansas
  - GSK Investigational Site, Topeka, Kansas
  - GSK Investigational Site, Fort Mitchell, Kentucky
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Madisonville, Kentucky
  - GSK Investigational Site, Paducah, Kentucky
  - GSK Investigational Site, Covington, Louisiana
  - GSK Investigational Site, Lake Charles, Louisiana
  - GSK Investigational Site, Shreveport, Louisiana
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Hyattsville, Maryland
  - GSK Investigational Site, Oxon Hill, Maryland
  - GSK Investigational Site, Haverhill, Massachusetts
  - GSK Investigational Site, Bay City, Michigan
  - GSK Investigational Site, Benzonia, Michigan
  - GSK Investigational Site, Bloomfield Hills, Michigan
  - GSK Investigational Site, Cadillac, Michigan
  - GSK Investigational Site, Dearborn, Michigan
  - GSK Investigational Site, Kalamazoo, Michigan
  - GSK Investigational Site, Saint Clair Shores, Michigan
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Gulfport, Mississippi
  - GSK Investigational Site, Picayune, Mississippi
  - GSK Investigational Site, Rolling Fork, Mississippi
  - GSK Investigational Site, Chesterfield, Missouri
  - GSK Investigational Site, Jefferson City, Missouri
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, Springfield, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, West Plains, Missouri
  - GSK Investigational Site, Billings, Montana
  - GSK Investigational Site, Butte, Montana
  - GSK Investigational Site, Great Falls, Montana
  - GSK Investigational Site, Broken Bow, Nebraska
  - GSK Investigational Site, Lincoln, Nebraska
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Berlin, New Jersey
  - GSK Investigational Site, Elizabeth, New Jersey
  - GSK Investigational Site, Haddon Heights, New Jersey
  - GSK Investigational Site, Hainesport, New Jersey
  - GSK Investigational Site, New Brunswick, New Jersey
  - GSK Investigational Site, Stratford, New Jersey
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, North Massapequa, New York
  - GSK Investigational Site, Asheboro, North Carolina
  - GSK Investigational Site, Asheville, North Carolina
  - GSK Investigational Site, Burlington, North Carolina
  - GSK Investigational Site, Calabash, North Carolina
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Fayetteville, North Carolina
  - GSK Investigational Site, Greensboro, North Carolina
  - GSK Investigational Site, Hickory, North Carolina
  - GSK Investigational Site, Huntersville, North Carolina
  - GSK Investigational Site, Lenoir, North Carolina
  - GSK Investigational Site, Mint Hill, North Carolina
  - GSK Investigational Site, Morehead City, North Carolina
  - GSK Investigational Site, Shelby, North Carolina
  - GSK Investigational Site, Tabor City, North Carolina
  - GSK Investigational Site, Akron, Ohio
  - GSK Investigational Site, Canal Fulton, Ohio
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Kettering, Ohio
  - GSK Investigational Site, Mason, Ohio
  - GSK Investigational Site, Maumee, Ohio
  - GSK Investigational Site, Thornville, Ohio
  - GSK Investigational Site, Zanesville, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Ashland, Oregon
  - GSK Investigational Site, Bensalem, Pennsylvania
  - GSK Investigational Site, Carlisle, Pennsylvania
  - GSK Investigational Site, Downington, Pennsylvania
  - GSK Investigational Site, Harrisburg, Pennsylvania
  - GSK Investigational Site, Landsdale, Pennsylvania
  - GSK Investigational Site, Melrose Park, Pennsylvania
  - GSK Investigational Site, Tipton, Pennsylvania
  - GSK Investigational Site, Uniontown, Pennsylvania
  - GSK Investigational Site, Cumberland, Rhode Island
  - GSK Investigational Site, East Providence, Rhode Island
  - GSK Investigational Site, Columbia, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Greer, South Carolina
  - GSK Investigational Site, Manning, South Carolina
  - GSK Investigational Site, Murrells Inlet, South Carolina
  - GSK Investigational Site, North Myrtle Beach, South Carolina
  - GSK Investigational Site, Orangeburg, South Carolina
  - GSK Investigational Site, Simpsonville, South Carolina
  - GSK Investigational Site, Taylors, South Carolina
  - GSK Investigational Site, Bristol, Tennessee
  - GSK Investigational Site, Chattanooga, Tennessee
  - GSK Investigational Site, Clarksville, Tennessee
  - GSK Investigational Site, Columbia, Tennessee
  - GSK Investigational Site, Fayetteville, Tennessee
  - GSK Investigational Site, Germantown, Tennessee
  - GSK Investigational Site, Johnson City, Tennessee
  - GSK Investigational Site, McKenzie, Tennessee
  - GSK Investigational Site, Memphis, Tennessee
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Tullahoma, Tennessee
  - GSK Investigational Site, Arlington, Texas
  - GSK Investigational Site, Bedford, Texas
  - GSK Investigational Site, Cleburne, Texas
  - GSK Investigational Site, Corpus Christi, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Deer Park, Texas
  - GSK Investigational Site, El Paso, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Hurst, Texas
  - GSK Investigational Site, Katy, Texas
  - GSK Investigational Site, Lake Jackson, Texas
  - GSK Investigational Site, Lewisville, Texas
  - GSK Investigational Site, Midland, Texas
  - GSK Investigational Site, North Richland Hills, Texas
  - GSK Investigational Site, Odessa, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Schertz, Texas
  - GSK Investigational Site, Sugar Land, Texas
  - GSK Investigational Site, Sugarland, Texas
  - GSK Investigational Site, Temple, Texas
  - GSK Investigational Site, Orem, Utah
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, West Jordan, Utah
  - GSK Investigational Site, West Valley City, Utah
  - GSK Investigational Site, South Burlington, Vermont
  - GSK Investigational Site, Burke, Virginia
  - GSK Investigational Site, Hampton, Virginia
  - GSK Investigational Site, Manassas, Virginia
  - GSK Investigational Site, Norfolk, Virginia
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Suffolk, Virginia
  - GSK Investigational Site, Virgina Beach, Virginia
  - GSK Investigational Site, Weber City, Virginia
  - GSK Investigational Site, Federal Way, Washington
  - GSK Investigational Site, Renton, Washington
  - GSK Investigational Site, Richland, Washington
  - GSK Investigational Site, Selah, Washington
  - GSK Investigational Site, Spokane, Washington
  - GSK Investigational Site, Tacoma, Washington
  - GSK Investigational Site, Lewisburg, West Virginia
  - GSK Investigational Site, Milwaukee, Wisconsin
- Germany (7):
  - GSK Investigational Site, Villingen-Schwenningen, Baden-Wurttemberg
  - GSK Investigational Site, Künzing, Bavaria
  - GSK Investigational Site, Kelkheim, Hesse
  - GSK Investigational Site, Rotenburg an der Fulda, Hesse
  - GSK Investigational Site, Bad Lauterberg im Harz, Lower Saxony
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Berlin, State of Berlin
- Hong Kong (4):
  - GSK Investigational Site, Chai Wan
  - GSK Investigational Site, Kwun Tong, Kowloon
  - GSK Investigational Site, Shatin
  - GSK Investigational Site, Tai Po
- India (4):
  - GSK Investigational Site, Aurangabad
  - GSK Investigational Site, Bangalore
  - GSK Investigational Site, Chennai
  - GSK Investigational Site, Pune
- Peru (3):
  - GSK Investigational Site, Ica, Ica
  - GSK Investigational Site, Lima, Lima Province
  - GSK Investigational Site, Callao, Lima
- Philippines (5):
  - GSK Investigational Site, Cebu City
  - GSK Investigational Site, Marikina City
  - GSK Investigational Site, Quezon City
  - GSK Investigational Site, San Juan City
  - GSK Investigational Site, Taytay Rizal
- Russia (2):
  - GSK Investigational Site, Smolensk
  - GSK Investigational Site, Yaroslavl
- Spain (5):
  - GSK Investigational Site, Alzira/Valencia
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Palma de Mallorca
  - GSK Investigational Site, Seville
- United Kingdom (4):
  - GSK Investigational Site, Blackpool, Lancashire
  - GSK Investigational Site, Coventry, West Midlands
  - GSK Investigational Site, Glasgow
  - GSK Investigational Site, London

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Home PD, Ahren B, Reusch JEB, Rendell M, Weissman PN, Cirkel DT, Miller D, Ambery P, Carr MC, Nauck MA. Three-year data from 5 HARMONY phase 3 clinical trials of albiglutide in type 2 diabetes mellitus: Long-term efficacy with or without rescue therapy. Diabetes Res Clin Pract. 2017 Sep;131:49-60. doi: 10.1016/j.diabres.2017.06.013. Epub 2017 Jun 15. PMID 28683300
- [Derived] Young MA, Wald JA, Matthews JE, Scott R, Hodge RJ, Zhi H, Reinhardt RR. Clinical pharmacology of albiglutide, a GLP-1 receptor agonist. Postgrad Med. 2014 Nov;126(7):84-97. doi: 10.3810/pgm.2014.11.2836. PMID 25387217
- [Derived] Young MA, Wald JA, Matthews JE, Yang F, Reinhardt RR. Effect of renal impairment on the pharmacokinetics, efficacy, and safety of albiglutide. Postgrad Med. 2014 May;126(3):35-46. doi: 10.3810/pgm.2014.05.2754. PMID 24918790
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 112757 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 112757 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 112757 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 112757 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 112757 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 112757 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 112757 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants (par.) who met eligibility criteria and completed a 6- to 8-week Run-in/Stabilization Period were then randomized to a 156-week Treatment Period, followed by 8 weeks of post-treatment follow-up. A total of 992 par. were screened; 685 par. were randomized, and 663 par. received >=1 treatment dose.
Groups:
- Placebo + Metformin + Glimepiride: Participants received albiglutide matching placebo as a subcutaneous injection weekly via a fully disposable pen injector system with open-label glimepiride (4 milligrams [mg] daily orally) with metformin (>=1500 mg daily orally). Participants did not receive investigational product during the Follow-up Period.
- Pioglitazone + Metformin + Glimepiride: Participants received pioglitazone (30 mg daily orally; with treatment-masked uptitration if needed to 45 mg) and albiglutide-matching placebo weekly as a subcutaneous injection via a fully disposable pen injector system with open-label glimepiride (4 mg daily orally) with metformin (>=1500 mg daily orally). Participants did not receive investigational product during the Follow-up Period.
- Albiglutide + Metformin + Glimepiride: Participants received pioglitazone-matching placebo daily orally and albiglutide (30 mg weekly; treatment-masked uptitration if needed to 50 mg weekly) as a subcutaneous injection via a fully disposable pen injector system with open-label glimepiride (4 mg daily orally) with metformin (>=1500 mg daily orally). Participants did not receive investigational product during the Follow-up Period.
Period: Treatment Period (TP) (156 Weeks)
Arm/Group | Placebo + Metformin + Glimepiride | Pioglitazone + Metformin + Glimepiride | Albiglutide + Metformin + Glimepiride
Started | 115 | 277 | 271
Completed | 55 | 159 | 152
Not Completed | 60 | 118 | 119
Not completed — Adverse Event | 11 | 29 | 22
Not completed — Protocol Violation | 4 | 7 | 1
Not completed — Noncompliance | 5 | 6 | 16
Not completed — Lost to Follow-up | 3 | 12 | 7
Not completed — Withdrawal by Subject | 32 | 46 | 64
Not completed — Physician Decision | 1 | 6 | 1
Not completed — Termination of Site by Sponsor | 3 | 8 | 5
Not completed — Missing | 0 | 1 | 0
Not completed — Persistant Elevated HbA1c Results | 0 | 0 | 1
Not completed — Pregnancy | 0 | 1 | 1
Not completed — Site Closed | 1 | 2 | 0
Not completed — Sponsor Decision on Blinding | 0 | 0 | 1
Period: Follow-up Period (FUP) (8 Weeks)
Arm/Group | Placebo + Metformin + Glimepiride | Pioglitazone + Metformin + Glimepiride | Albiglutide + Metformin + Glimepiride
Started | 114 (Par. withdrawing from the TP could enter the FUP. One par. did not participate in the FUP.) | 273 (Par. withdrawing from the TP could enter the FUP. Four par. did not participate in the FUP.) | 266 (Par. withdrawing from the TP could enter the FUP. Five par. did not participate in the FUP.)
Completed | 86 | 217 | 204
Not Completed | 28 | 56 | 62
Not completed — Adverse Event | 1 | 2 | 1
Not completed — Noncompliance | 1 | 0 | 5
Not completed — Lost to Follow-up | 8 | 20 | 29
Not completed — Withdrawal by Subject | 12 | 21 | 19
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Termination of Study by Sponsor | 3 | 10 | 5
Not completed — Informed Consent Recalled by Participant | 1 | 0 | 0
Not completed — Investigator Closed Study at Site | 1 | 0 | 0
Not completed — Site Closed | 0 | 1 | 0
Not completed — Site Closing and Withdrew Consent | 1 | 0 | 1
Not completed — Unable to Complete Follow-up | 0 | 1 | 0
Not completed — Missing Follow-up Status | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo + Metformin + Glimepiride | Pioglitazone + Metformin + Glimepiride | Albiglutide + Metformin + Glimepiride | Total
Number analyzed (Participants) | 115 | 277 | 271 | 663
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.7 (9.59) | 55.7 (9.39) | 54.5 (9.47) | 55.2 (9.46)
Gender [Count of Participants; unit: Participants]
  Female | 45 | 129 | 136 | 310
  Male | 70 | 148 | 135 | 353
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 10 | 24 | 34 | 68
  American Indian or Alaskan Native | 9 | 10 | 22 | 41
  Asian - Central/South Asian Heritage | 6 | 6 | 8 | 20
  Asian - East Asian Heritage | 2 | 8 | 12 | 22
  Asian - Japanese Heritage | 0 | 1 | 2 | 3
  Asian - South East Asian Heritage | 7 | 24 | 14 | 45
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 0 | 2
  White - Arabic/North African Heritage | 1 | 2 | 2 | 5
  White - White/Caucasian/European Heritage | 79 | 201 | 176 | 456
  Mexican American | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (BL) in Glycosylated Hemoglobin (HbA1c) at Week 52
Description: HbA1c is a form of hemoglobin that is measured primarily to identify the average plasma glucose concentration over a 2- to 3-month period. The BL HbA1c value is defined as the last non-missing value before the start of treatment. Change from BL was calculated as the value at Week 52 minus the value at BL. Based on analysis of covariance (ANCOVA): change = treatment + BL HbA1c + prior myocardial infarction history + age category + region. The last observation carried forward (LOCF) method was used to impute missing post-BL HbA1c values; the last non-missing post-BL on-treatment measurement was used to impute the missing measurement. HbA1c values obtained after hyperglycemic rescue were treated as missing and were replaced with pre-rescue values. Nine par. with post-BL values obtained >14 days after the last dose or after hyperglycemic rescue were included in the analysis population but were not analyzed for this endpoint.
Time Frame: Baseline and Week 52
Population: Intent-to-Treat (ITT) Population with LOCF: all randomized par. who received >=1 dose of study medication and who had a BL assessment and >=1 post-BL assessment of HbA1c. Only par. with a value at BL and at the specified visit were analyzed. Values were carried forward for par. who were rescued or discontinued from active treatment before Week 52.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c in the blood
Arm/Group | Placebo + Metformin + Glimepiride | Pioglitazone + Metformin + Glimepiride | Albiglutide + Metformin + Glimepiride
Number analyzed (Participants) | 115 | 268 | 265
Percentage of HbA1c in the blood | 0.33 (0.083) | -0.80 (0.055) | -0.55 (0.055)
Statistical Analysis 1: Comparison: Placebo + Metformin + Glimepiride vs Albiglutide + Metformin + Glimepiride; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = -0.87, 95% CI 2-sided [-1.07 to -0.68]
Statistical Analysis 2: Comparison: Pioglitazone + Metformin + Glimepiride vs Albiglutide + Metformin + Glimepiride; Test type: Non-Inferiority or Equivalence — The p-value is from a one-sided t-test testing at the 0.025 level of significance whether or not the difference of least square means (albiglutide - pioglitazone) is less than or equal to the pre-specified non-inferiority margin of 0.3%; p = 0.2685, t-test, 1 sided; Mean Difference (Net) = 0.25, 95% CI 2-sided [0.10 to 0.40]

2. Secondary Outcome: Change From Baseline in HbA1c at Week 104 and Week 156
Description: HbA1c is a form of hemoglobin that is measured primarily to identify the average plasma glucose concentration over a 2- to 3-month period. The Baseline HbA1c value is defined as the last non-missing value before the start of treatment. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. This analysis used observed HbA1c values, excluding those obtained after hyperglycemia rescue; no missing data imputation was performed.
Time Frame: Baseline, Week 104, and Week 156
Population: ITT Population with observed values. Only those participants with a value at Baseline and at the specified visit were analyzed (represented by n=X, X, X in the category titles).
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c in the blood
Arm/Group | Placebo + Metformin + Glimepiride | Pioglitazone + Metformin + Glimepiride | Albiglutide + Metformin + Glimepiride
Number analyzed (Participants) | 12 | 130 | 104
Percentage of HbA1c in the blood
  Week 104, n=12, 130, 104 | -0.32 (0.552) | -1.09 (1.119) | -0.76 (1.009)
  Week 156, n=9, 89, 71 | -0.10 (0.923) | -0.97 (1.063) | -0.46 (1.113)

3. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 52
Description: The FPG test measures blood sugar levels after the participant has not eaten (fasted) for 12 to 14 hours. The Baseline FPG value is the last non-missing value before the start of treatment. The LOCF method was used to impute missing post-Baseline FPG values. FPG values obtained after hyperglycemia rescue were treated as missing and replaced with pre-rescue values. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. Based on ANCOVA: change = treatment + Baseline FPG + Baseline HbA1c category + prior myocardial infarction history + age category + region.
Time Frame: Baseline and Week 52
Population: Intent-to-Treat (ITT) Population with LOCF. Only those participants with a value at Baseline and at the specified visit were analyzed. Values were carried forward for participants who were rescued or discontinued from active treatment before Week 52.
Measure: Least Squares Mean (Standard Error); unit: Millimoles per liter (mmol/L)
Arm/Group | Placebo + Metformin + Glimepiride | Pioglitazone + Metformin + Glimepiride | Albiglutide + Metformin + Glimepiride
Number analyzed (Participants) | 115 | 272 | 268
Millimoles per liter (mmol/L) | 0.64 (0.243) | -1.74 (0.158) | -0.69 (0.159)

4. Secondary Outcome: Change From Baseline in FPG at Week 104 and Week 156
Description: The FPG test measures blood sugar levels after the participant has not eaten (fasted) for 12 to 14 hours. The Baseline FPG value is the last non-missing value before the start of treatment. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. This analysis used observed FPG values excluding those obtained after hyperglycemia rescue; no missing data imputation was performed.
Time Frame: Baseline, Week 104, and Week 156
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Placebo + Metformin + Glimepiride | Pioglitazone + Metformin + Glimepiride | Albiglutide + Metformin + Glimepiride
Number analyzed (Participants) | 12 | 128 | 103
Millimoles per liter (mmol/L)
  Week 104, n=12, 128, 103 | 0.43 (3.346) | -1.98 (3.471) | -0.99 (3.083)
  Week 156, n=9, 88, 71 | -0.50 (4.093) | -1.94 (3.127) | -0.88 (2.652)

5. Secondary Outcome: Time to Hyperglycemia Rescue
Description: Participants who experienced persistent hyperglycemia (high blood glucose) could have qualified for hyperglycemia rescue. The conditions for hyperglycemia rescue were as follows: FPG >=280 milligrams/deciliter (mg/dL) between >=Week 2 and <Week 4; FPG >=250 mg/dL between >=Week 4 and <Week 12; HbA1c >=8.5% and a <=0.5% reduction from Baseline between >=Week 12 and <Week 24; HbA1c >=8.5% between >=Week 24 and <Week 48; HbA1c >=8.0% between >= Week 48 and <Week 156. Participants could have been rescued at any time on or after Week 2. Time to hyperglycemia rescue is defined as the time between the date of the first dose of study medication and the date of hyperglycemia rescue plus 1 day, or the time between the date of the first dose of study medication and the date of the last visit during the active treatment period plus 1 day for participants not requiring rescue. This time was divided by 7 to express the result in weeks.
Time Frame: From the start of study medication until the end of the treatment (up to Week 156)
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Placebo + Metformin + Glimepiride | Pioglitazone + Metformin + Glimepiride | Albiglutide + Metformin + Glimepiride
Number analyzed (Participants) | 115 | 273 | 269
Weeks | 49.57 [38.86 to 55.14] | NA [NA to NA] — There were too few events of hyperglycemia rescue (<50% of participants with events) to calculate the median and confidence interval. | 137.71 [93.71 to NA] — The upper bound of the 95% confidence interval is not available because it is beyond the study duration.

6. Secondary Outcome: Number of Participants Who Achieved Clinically Meaningful HbA1c Response Levels of <6.5%, <7%, and <7.5% at Week 52
Description: The number of participants who acheieved the HbA1c treatment goal (i.e., HbA1c response levels of <6.5%, <7%, and <7.5% at Week 52) was assessed. Values were carried forward for participants who were rescued or discontinued from active treatment before Week 52.
Time Frame: Week 52
Population: ITT Population with LOCF. Only those participants with a value at Baseline and at the specified visit were analyzed.
Measure: Number; unit: Participants
Arm/Group | Placebo + Metformin + Glimepiride | Pioglitazone + Metformin + Glimepiride | Albiglutide + Metformin + Glimepiride
Number analyzed (Participants) | 115 | 268 | 265
Participants
  HbA1c <6.5% | 4 | 37 | 27
  HbA1c <7.0% | 10 | 94 | 79
  HbA1c <7.5% | 19 | 150 | 126

7. Secondary Outcome: Number of Participants Who Achieved Clinically Meaningful HbA1c Response Levels of <6.5%, <7%, and <7.5% at Week 156
Description: The number of participants who acheieved the HbA1c treatment goal (i.e., HbA1c response levels of <6.5%, <7%, and <7.5% at Week 156) was assessed.
Time Frame: Week 156
Population: ITT Population with observed values. Only those participants with a value at Baseline and at the specified visit were analyzed. This analysis used observed HbA1c values excluding those obtained after hyperglycemia rescue; no missing data imputation was performed.
Measure: Number; unit: Participants
Arm/Group | Placebo + Metformin + Glimepiride | Pioglitazone + Metformin + Glimepiride | Albiglutide + Metformin + Glimepiride
Number analyzed (Participants) | 9 | 89 | 71
Participants
  HbA1c <6.5% | 1 | 23 | 16
  HbA1c <7.0% | 3 | 44 | 26
  HbA1c <7.5% | 5 | 68 | 45

8. Secondary Outcome: Change From Baseline in Body Weight at Week 52
Description: The Baseline value is the last non-missing value before the start of treatment. Change from Baseline was calculated as the post-Baseline weight minus the Baseline weight. The LOCF method was used to impute missing post-Baseline weight values. Weight values obtained after hyperglycemia rescue were treated as missing and replaced with pre-rescue values. Based on ANCOVA: change = treatment + Baseline weight + Baseline HbA1c category + prior myocardial infarction history + age category + region.
Time Frame: Baseline and Week 52
Population: ITT Population with LOCF. Only those participants with a value at Baseline and at the specified visit were analyzed. Values were carried forward for participants who were rescued or discontinued from active treatment before Week 52.
Measure: Least Squares Mean (Standard Error); unit: Kilograms
Arm/Group | Placebo + Metformin + Glimepiride | Pioglitazone + Metformin + Glimepiride | Albiglutide + Metformin + Glimepiride
Number analyzed (Participants) | 115 | 272 | 268
Kilograms | -0.40 (0.362) | 4.43 (0.235) | -0.42 (0.237)

9. Secondary Outcome: Change From Baseline in Body Weight at Week 104 and Week 156
Description: The Baseline value is the last non-missing value before the start of treatment. Change from Baseline was calculated as the post-Baseline weight minus the Baseline weight. This analysis used observed body weight values excluding those obtained after hyperglycemia rescue; no missing data imputation was performed.
Time Frame: Baseline, Week 104, and Week 156
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Placebo + Metformin + Glimepiride | Pioglitazone + Metformin + Glimepiride | Albiglutide + Metformin + Glimepiride
Number analyzed (Participants) | 12 | 130 | 104
Kilograms
  Week 104, n=12, 130, 104 | -2.16 (3.603) | 6.28 (6.189) | -0.90 (3.721)
  Week 156, n=9, 90, 71 | -4.47 (5.380) | 6.52 (6.332) | -1.53 (3.880)

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious AEs, defined as those events that had a start date on or after the first day of study medication and within 56 days after the end of study medication (up to Week 156), are reported.
Description: SAEs and non-serious AEs are reported for members of the Safety Population, comprised of all participants who received at least one dose of study treatment.
Arm/Group | Placebo + Metformin + Glimepiride | Pioglitazone + Metformin + Glimepiride | Albiglutide + Metformin + Glimepiride
Serious Adverse Events (participants affected / at risk) | 21/115 | 48/277 | 39/271
Other Adverse Events (participants affected / at risk) | 81/115 | 228/277 | 228/271
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Metformin + Glimepiride (N=115) | Pioglitazone + Metformin + Glimepiride (N=277) | Albiglutide + Metformin + Glimepiride (N=271)
Coronary artery disease (Cardiac disorders) | 0 | 4 | 3
Cardiac failure congestive (Cardiac disorders) | 1 | 4 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 3
Acute myocardial infarction (Cardiac disorders) | 1 | 2 | 0
Sick sinus syndrome (Cardiac disorders) | 0 | 1 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0
Arteriosclerosis coronary (Cardiac disorders) | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 2 | 1 | 2
Cellulitis (Infections and infestations) | 2 | 1 | 0
Diabetic foot infection (Infections and infestations) | 1 | 0 | 1
Abscess (Infections and infestations) | 0 | 1 | 0
Febrile infection (Infections and infestations) | 1 | 0 | 0
Gangrene (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0
Infected bites (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 1 | 0 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0 | 0
Localised infection (Infections and infestations) | 0 | 1 | 0
Meningitis pneumococcal (Infections and infestations) | 1 | 0 | 0
Pancreatitis viral (Infections and infestations) | 0 | 0 | 1
Peritonitis (Infections and infestations) | 0 | 1 | 0
Postoperative wound infection (Infections and infestations) | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0
Tracheobronchitis (Infections and infestations) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 3 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 2 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 2 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Hypertensive encephalopathy (Nervous system disorders) | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0
Metabolic encephalopathy (Nervous system disorders) | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0
Myelitis transverse (Nervous system disorders) | 0 | 0 | 1
Nerve compression (Nervous system disorders) | 0 | 1 | 0
Trigeminal neuralgia (Nervous system disorders) | 0 | 1 | 0
Vith nerve paralysis (Nervous system disorders) | 0 | 1 | 0
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 2
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Sigmoiditis (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Chest pain (General disorders) | 1 | 4 | 2
Sudden death (General disorders) | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 2 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Bipolar disorder (Psychiatric disorders) | 0 | 0 | 1
Major depression (Psychiatric disorders) | 0 | 1 | 0
Panic disorder (Psychiatric disorders) | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 3 | 0 | 0
Glomerulonephritis acute (Renal and urinary disorders) | 1 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 2
Peripheral artery stenosis (Vascular disorders) | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Metformin + Glimepiride (N=115) | Pioglitazone + Metformin + Glimepiride (N=277) | Albiglutide + Metformin + Glimepiride (N=271)
Nasopharyngitis (Infections and infestations) | 16 | 28 | 43
Upper respiratory tract infection (Infections and infestations) | 21 | 50 | 34
Urinary tract infection (Infections and infestations) | 9 | 31 | 24
Sinusitis (Infections and infestations) | 7 | 16 | 18
Bronchitis (Infections and infestations) | 7 | 25 | 16
Influenza (Infections and infestations) | 5 | 10 | 16
Gastroenteritis (Infections and infestations) | 5 | 10 | 9
Pharyngitis (Infections and infestations) | 5 | 9 | 8
Gastroenteritis viral (Infections and infestations) | 2 | 3 | 6
Furuncle (Infections and infestations) | 0 | 2 | 6
Tooth abscess (Infections and infestations) | 4 | 3 | 5
Herpes zoster (Infections and infestations) | 3 | 1 | 4
Cellulitis (Infections and infestations) | 2 | 13 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 28 | 115 | 84
Dyslipidaemia (Metabolism and nutrition disorders) | 1 | 4 | 7
Decreased appetite (Metabolism and nutrition disorders) | 3 | 3 | 5
Hyperlipidaemia (Metabolism and nutrition disorders) | 3 | 4 | 4
Diarrhoea (Gastrointestinal disorders) | 12 | 23 | 37
Nausea (Gastrointestinal disorders) | 7 | 20 | 30
Abdominal pain (Gastrointestinal disorders) | 2 | 7 | 17
Constipation (Gastrointestinal disorders) | 7 | 11 | 14
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 9 | 12
Dyspepsia (Gastrointestinal disorders) | 1 | 2 | 10
Vomiting (Gastrointestinal disorders) | 4 | 14 | 6
Abdominal pain upper (Gastrointestinal disorders) | 1 | 7 | 6
Gastritis (Gastrointestinal disorders) | 3 | 5 | 5
Toothache (Gastrointestinal disorders) | 1 | 9 | 4
Abdominal distension (Gastrointestinal disorders) | 3 | 4 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 23 | 26
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 24 | 24
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 14 | 12
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 7 | 12
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 | 12 | 11
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 11 | 8
Tendonitis (Musculoskeletal and connective tissue disorders) | 3 | 4 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 8 | 4
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 | 4 | 2
Injection site reaction (General disorders) | 1 | 8 | 32
Oedema peripheral (General disorders) | 9 | 41 | 12
Fatigue (General disorders) | 6 | 15 | 8
Chest pain (General disorders) | 3 | 4 | 2
Oedema (General disorders) | 0 | 8 | 1
Headache (Nervous system disorders) | 6 | 25 | 21
Dizziness (Nervous system disorders) | 6 | 9 | 16
Neuropathy peripheral (Nervous system disorders) | 1 | 12 | 13
Hypoaesthesia (Nervous system disorders) | 1 | 7 | 7
Diabetic neuropathy (Nervous system disorders) | 4 | 4 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 19 | 28
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 9 | 5
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 6 | 2
Ligament sprain (Injury, poisoning and procedural complications) | 2 | 4 | 8
Contusion (Injury, poisoning and procedural complications) | 5 | 8 | 7
Muscle strain (Injury, poisoning and procedural complications) | 5 | 6 | 7
Excoriation (Injury, poisoning and procedural complications) | 6 | 7 | 4
Procedural pain (Injury, poisoning and procedural complications) | 1 | 8 | 3
Rib Fracture (Injury, poisoning and procedural complications) | 3 | 1 | 2
Hypertension (Vascular disorders) | 11 | 27 | 22
Diabetic retinopathy (Eye disorders) | 3 | 17 | 10
Cataract (Eye disorders) | 3 | 13 | 8
Insomnia (Psychiatric disorders) | 2 | 9 | 11
Anxiety (Psychiatric disorders) | 1 | 7 | 9
Depression (Psychiatric disorders) | 3 | 12 | 5
Cardiac murmur (Investigations) | 0 | 3 | 6
Gamma-glutamyltransferase increased (Investigations) | 1 | 1 | 6
Blood creatinine increased (Investigations) | 1 | 6 | 1
Weight increased (Investigations) | 0 | 21 | 0
Anaemia (Blood and lymphatic system disorders) | 4 | 24 | 13
Leukocytosis (Blood and lymphatic system disorders) | 3 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 4 | 9 | 5
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 1 | 6 | 2
Dry Skin (Skin and subcutaneous tissue disorders) | 3 | 2 | 2
Vertigo (Ear and labyrinth disorders) | 1 | 7 | 9
Seasonal allergy (Immune system disorders) | 3 | 4 | 5
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 4 | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.